CLINICAL TRIAL: NCT04599868
Title: High Versus Low Dose of Magnesium Sulfate as Initial Tocolytic Agent for Preterm Labour in Symptomatic Placenta Previa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa M. Mostafa, Resident of obstetrics &Gynecology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mgso4 for PTL in pp
Record Dates: First submitted 2020-10-05; First posted 2020-10-23 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Placenta Previa Bleeding
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose of magnesium sulfate group (Active Comparator): patients will receive 4 g intravenous loading dose of magnesium sulfate on 150 ml saline over 20 minute period. Patients then will receive maintenance therapy with magnesium sulfate 1g / h
  Interventions: Drug: Magnesium sulfate
- High dose of magnesium sulfate group (Active Comparator): patients will receive 4 g intravenous loading dose of magnesium sulfate on 150 ml saline over 20 minute period. Patients then will receive maintenance therapy with magnesium sulfate 2g/h
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — Patients will be assessed hourly for pulse and blood pressure, contraction frequency, vaginal bleeding. With strict monitoring for symptoms of magnesium sulfate toxicity.
  All patients will receive dexamethasone to enhance fetal lung maturity. Rhesus factor status will be determined for all patients, . Hb level will be measured and anemic patients will receive correction by blood transfusion Cervical length will be measured after 24 h& 48 h from administration of magnesium sulfate in both groups Maternal serum magnesium will be measured at admission and after 4 hours ,12 hours and 24 hours after administration of magnesium sulfate Patients of both groups will be assessed for their neonatal outcomes include deaths and gestational age at delivery, fetal birth weight. Apgar score at five minutes, neonatal intensive care unit admission and duration of admission and neonatal calcium level at time of delivery will be also assessed.

SUMMARY:
To assess the efficacy and safety of alternative magnesium sulfate regimens when used as single agent tocolytic therapy for prevention of preterm labour in patients with symptomatic placenta previa and subsequent changes in the cervical length .

DETAILED DESCRIPTION:
Placenta previa is implantation of placenta on or near internal os .It is classified into major degree when lower edge of placenta lies within 2 cm from internal os , and minor degree if lower edge of placenta at lower uterine segment but more than 2 cm from internal os .

There are many risk factors for developing placenta previa including multi parity , multiple pregnancy , increased maternal age (>35y ) , previous uterine surgery , history of placenta previa (4-8%) .

A significant degree of uterine contractility has been observed with symptomatic placenta previa. It is directly associated with vaginal bleeding. However, a large percentage of women who have placenta previa associated with haemorrhage will experience subclinical uterine contractions before the onset of overt vaginal bleeding. Therefore, the use of tocolytic agents in management of placenta previa seems reasonable .

Magnesium sulfate alters calcium up take, binding and distribution in smooth muscles of the uterus, so reduces the frequency of cell depolarization and inhibits myometrial contraction .

In addition to its tocolytic action magnesium sulfate also provide neuroprotection to preterm infant . .

At women Health Hospital, Assiut University, Egypt our policy is using magnesium sulfate as first line for tocolysis for placenta previa patients with preterm uterine contractions. By giving a loading dose of 4 g on 150 ml saline intravenous infusion over 20 minutes, and a maintenance dose of 6g/6h on 500 ml saline slow intra venous infusion

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy.
2. Gestational age between 28 weeks to 37 weeks.
3. Patients presented to the hospital with per vaginal bleeding and in whom a clinical diagnosis of placenta previa is confirmed by trans vaginal ultrasound.
4. Placenta previa with preterm uterine contractions (< 3 contractions in 10 minutes)
5. Ability to provide informed consent.

Exclusion Criteria:

1. Placental abruption .
2. Women with placenta previa and severe attack of bleeding need immediate termination
3. Clinical criteria of intra uterine infection.
4. intrauterine growth restriction .
5. Fetal anomalies.
6. Fetal distress.
7. intrauterine fetal death.
8. Preterm rupture of membrane
9. High order multiple pregnancies.
10. Treatment with any tocolytic agent before maternal transport.
11. Inability or refusal to provide informed consent.
12. Women with any contraindication for use of magnesium sulfate as patients with renal failure.
13. Patients with bleeding disorder or on anticoagulant therapy .

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — only females
Enrollment: 130 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy (postponing delivery for 48h - till administration of dexamethasone ) of different regimens 0f MgSO4 in patients with pp in preterm . 2) Different regimens of MGSO4 and changes in cervical length | 48 hour
  comparing efficacy of low vs high dose of MgSO4 to postpone preterm delivery in patients with symptomatic pp and subsequent changes in cervical length

SECONDARY OUTCOMES:
Gestational age at delivery | at time of delivery
birth weight | at time of delivery
number of full term babies | at time of delivery
fetal and Neonatal death . | at time of delivery
Apgar score at five minutes . | 5 minutes
Neonatal intensive care unit admission & duration of admission | at time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morfaw F, Fundoh M, Bartoszko J, Mbuagbaw L, Thabane L. Using tocolysis in pregnant women with symptomatic placenta praevia does not significantly improve prenatal, perinatal, neonatal and maternal outcomes: a systematic review and meta-analysis. Syst Rev. 2018 Dec 27;7(1):249. doi: 10.1186/s13643-018-0923-2. PMID 30591076
- [Background] Marshall NE, Fu R, Guise JM. Impact of multiple cesarean deliveries on maternal morbidity: a systematic review. Am J Obstet Gynecol. 2011 Sep;205(3):262.e1-8. doi: 10.1016/j.ajog.2011.06.035. Epub 2011 Jun 15. PMID 22071057
- [Background] Milosevic J, Lilic V, Tasic M, Radovic-Janosevic D, Stefanovic M, Antic V. [Placental complications after a previous cesarean section]. Med Pregl. 2009 May-Jun;62(5-6):212-6. doi: 10.2298/mpns0906212m. Serbian. PMID 19650556
- [Background] Wennberg AL, Opdahl S, Bergh C, Aaris Henningsen AK, Gissler M, Romundstad LB, Pinborg A, Tiitinen A, Skjaerven R, Wennerholm UB. Effect of maternal age on maternal and neonatal outcomes after assisted reproductive technology. Fertil Steril. 2016 Oct;106(5):1142-1149.e14. doi: 10.1016/j.fertnstert.2016.06.021. Epub 2016 Jul 9. PMID 27399261
- [Background] Saleh Gargari S, Seify Z, Haghighi L, Khoshnood Shariati M, Mirzamoradi M. Risk Factors and Consequent Outcomes of Placenta Previa: Report From a Referral Center. Acta Med Iran. 2016 Nov;54(11):713-717. PMID 28033694
- [Background] ) Almnabri, A.A., et al., Management of Placenta Previa During Pregnancy. The Egyptian Journal of Hospital Medicine, 2017. 68(3): p. 1549-1553
- [Background] Sharma A, Suri V, Gupta I. Tocolytic therapy in conservative management of symptomatic placenta previa. Int J Gynaecol Obstet. 2004 Feb;84(2):109-13. doi: 10.1016/S0020-7292(03)00198-X. PMID 14871511
- [Background] McNamara HC, Crowther CA, Brown J. Different treatment regimens of magnesium sulphate for tocolysis in women in preterm labour. Cochrane Database Syst Rev. 2015 Dec 14;2015(12):CD011200. doi: 10.1002/14651858.CD011200.pub2. PMID 26662716
- [Background] Kawagoe Y, Sameshima H, Ikenoue T, Yasuhi I, Kawarabayashi T. Magnesium sulfate as a second-line tocolytic agent for preterm labor: a randomized controlled trial in Kyushu Island. J Pregnancy. 2011;2011:965060. doi: 10.1155/2011/965060. Epub 2011 Jun 16. PMID 21773032